CLINICAL TRIAL: NCT06095427
Title: A Randomized, Double Blind, Three-Arm, Parallel Group, Pharmacokinetic Similarity Study in Healthy Male Subjects to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of LY06006 Versus US Prolia and EU Prolia by Single-Dose Subcutaneous Injection
Brief Title: A Pharmacokinetic Similarity Study in Healthy Male Subjects to Evaluate Pharmacokinetics, Pharmacodynamics, Safety and Immunogenicity of LY06006 Versus US-Prolia and EU-Prolia by Single-dose Subcutaneous Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LY06006/CT-EUR-101; 247228 (Other: CRO); 2020-000286-16 (EudraCT Number)
Record Dates: First submitted 2023-05-05; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, double-blind, single-dose, three-arm, parallel-group study designed to demonstrate the PK similarity between LY06006, US-Prolia and EU-Prolia and to evaluate the safety, tolerability, immunogenicity and PD of LY06006 compared with US-Prolia and EU-Prolia.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LY06006 (Experimental): 60 mg LY006006
  Interventions: Biological: LY06006 (Denosumab Biosimilar)
- US-Prolia (Active Comparator): 60 mg US-Prolia
  Interventions: Biological: US-Prolia (Denosumab)
- EU-Prolia (Active Comparator): 60 mg EU-Prolia
  Interventions: Biological: EU-Prolia

INTERVENTIONS:
Biological: LY06006 (Denosumab Biosimilar) — single dose of 60 mg LY006006 s.c.
  Arms: LY06006
Biological: US-Prolia (Denosumab) — single dose of 60 mg US-Prolia s.c.
  Arms: US-Prolia
Biological: EU-Prolia — single dose of 60 mg EU-Prolia s.c.
  Arms: EU-Prolia

SUMMARY:
This trial is a randomized, double-blind, three-arm, parallel-group, pharmacokinetic study. The purpose of this study is to demonstrate pharmacokinetic (PK) similarity and to compare safety, immunogenicity and pharmacodynamics (PD) between the test product L06006 and the reference products US-Prolia and EU-Prolia in healthy male subjects. A total of 300 healthy male subjects aged 28 to 65 years (both inclusive) will be randomized 1:1:1 to receive a single subcutaneous (s.c.) injection of either LY06006 or US-Prolia or EU-Prolia on Day 1 and then be followed for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males aged 28 - 65 years, both inclusive;
2. Body mass index (BMI) between 18 to < 30 kg/m2 and body weight of 60 - 90 kg (both inclusive);
3. Subjects must give written informed consent before any assessment is performed and has to understand the study and must be willing to follow and complete all the test procedures;
4. Clinically acceptable physical exams and laboratory tests (blood hematology, blood chemistry, coagulation, urinalysis) and no history or evidence of any clinically significant medical disorder that would pose a risk to subject safety or interfere with study evaluations or procedures;
5. Available for long term clinical assessments (36 weeks post-dose) for PK/PD and immunogenicity assessments;
6. Subjects and their female partners who are of childbearing potential must be using 2 forms of birth control (1 of which is a highly effective method† and 1 must be a barrier method‡) or abstain from sexual intercourse with a female partner (acceptable only if it is the subject's usual form of birth control/lifestyle choice) starting at Day -1 and throughout the study period and for at least 1 month after the end of EoS Visit. A condom is required to be used also by vasectomized men to prevent delivery of the drug via seminal fluid.

Highly effective forms of birth control include (i.e., less than 1% failure rate per year when used consistently and correctly):

* hormonal contraception, i.e., oral, injectable or implantable hormonal contraceptives for the female partner (Note: Not all oral contraception methods have a low failure rate.).
* hormonal or non-hormonal intrauterine device (IUD), established IUD (loop) or intrauterine system for the female partner.
* the subject has undergone effective surgical sterilization before he entered the study.
* the subject's female partner has undergone effective surgical sterilization before the subject entered the clinical trial and she is the sole sexual partner of the subject during the study.

Acceptable methods of surgical sterilization are:

* Surgical bilateral oophorectomy for the female partner (with or without hysterectomy) at least 6 weeks before the SCR Visit.
* Hysterectomy for the female partner at least 6 weeks before the SCR Visit.
* Bilateral tubal ligation for the female partner at least 6 weeks before the SCR Visit.

Barrier methods of birth control:

* Condom without spermicidal foam / gel / film / cream / suppository or fat- or oil-containing lubricant.
* Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam / gel / film / cream / suppository for the female partner.

Exclusion Criteria:

1. Subjects with prior exposure to denosumab (Prolia, Xgeva, or biosimilar denosumab);
2. Use of any other monoclonal antibodies or fusion proteins within the 3 months or 5 half-lives (whatever is longer) before the date of administration of the IMP;
3. Subjects being on a special diet or with significant weight loss from a weight reduction diet (e.g., more than approx. 5 kg within 1 month) before the SCR Visit or unwilling to maintain the same weight for the duration of the study;
4. Donation or loss of ≥ 500 mL of blood within 8 weeks prior to dosing, or longer if required by local regulation. Plasma donation within 28 days prior to dosing;
5. Diseases and conditions that affect bone metabolism e.g., osteoporosis, hypo/hyper-parathyroidism (excluding isolated deviations of parathormone assessed as not clinically significant); hypo-/hyperthyroidism, Cushing's syndrome, malabsorption syndromes, rheumatoid arthritis, psoriatic arthritis, osteomalacia, bone fractures within 6 months, or any contraindications to denosumab therapy;
6. Vitamin D deficiency (serum 25-hydroxy vitamin D < 20 ng/mL). For subjects with vitamin D deficiency, a single attempt at oral replenishment with re-evaluation prior to randomization is permitted (see Section 5.5);
7. Subjects with systolic blood pressure (SBP) ≥ 140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg and / or pulse < 50 or > 90 bpm (mean of triplicate measurements. Subjects with pulse rate between 45 and 50 bpm (inclusive) may be enrolled provided they have a normal thyroid function, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia (e.g., cardiovascular disease);
8. Subjects with abnormal ECGs (QTcF > 450 ms, signs of ischemia, sinus tachycardia [heart rate, HR > 90] or sinus bradycardia [HR < 50], ventricular conduct delay [QRS > 120 ms] or others) which, in the judgment of the Investigator or any of the Sub-Investigators, may be clinically relevant. Subjects with heart rate between 45 and 50 bpm (inclusive) may be enrolled provided they have a normal thyroid function, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia (e.g., cardiovascular disease). Potential cardiovascular disease resulting in bradycardia should be excluded by further investigations on the discretion of the Investigator;
9. Any clinically relevant laboratory findings that, in the opinion of the Investigator, would preclude inclusion in the trial; subjects with creatinine above Upper Limit of Normal (ULN) or liver enzymes (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) 1.5-fold above ULN will be excluded;
10. Subject presents with any psychiatric disorder, which may prevent the subject from completing the study or interfere with the interpretation of the study results;
11. Subjects with current or a history of clinically significant (or "serious") skin infections or skin disorders;
12. Subject has a history or presence of anemia or coagulopathy;
13. Significant changes in physical activity during the 6 months before IMP administration or constant levels of intense physical exercise;
14. Positive test results for hepatitis B surface antigen (HbsAg), anti-hepatitis B core (anti-HBc) antibodies indicative of active hepatitis, optionally Hepatitis B surface antibody (anti-HBS), hepatitis A virus antibodies (immunoglobulin M [IgM]), hepatitis C virus (HCV) antibodies and / or human immunodeficiency virus (HIV) type-1 and / or type-2 antibodies at the SCR Visit;
15. Use of any prescription drug or any over-the-counter (OTC) drug within the 2 weeks (or less than 5 x the half-life of that medication, whichever is longer) including herbal supplements, or prescribed/ non-prescribed marijuana derivatives before the date of administration of the IMP (excluding localized use not intended to have systemic action and occasional use of paracetamol of up to 2 g per day), which, in the judgment of the Investigator or Sub-Investigators, may affect participation in this clinical study. Vitamins, minerals and nutritional supplements may be taken at the discretion of the Investigator;
16. Prior use of any medications that may affect bone turnover within 12 months of IMP administration and for the duration of the study. This includes medications such as, but not limited to: bisphosphonates, fluoride, or selective estrogen receptor modulator, such as ralaxofene, calcitonin, strontium, parathyroid hormone or derivatives, supplemental vitamin D [> 1000 IU/day], except for the potential vitamin D replenishment after SCR, glucocorticosteroids, anabolic steroids, calcitriol, diuretics. Current use of anti-angiogenic drugs;
17. Receiving or has received any investigational drug (or is currently using an investigational device) within 60 days before receiving IMP, or at least 10 times the respective elimination half-life (whichever period is longer) and for the duration of the study;
18. Men with partners who are pregnant or planning to become pregnant while the subject is on study until through at least 1 month after the end of the study;
19. Intent to donate sperm during the study through at least 1 month after the end of the study;
20. Unwilling or unable to limit alcohol consumption throughout the course of the study. Alcohol is prohibited 24 hours prior to each visit in the clinical and throughout confinement. Alcohol is also limited to no more than 168 g pure alcohol per week (10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) during the outpatient period.;
21. Positive urine screen for alcohol and/or drugs with a high potential for abuse at SCR or Day -1;
22. Any other condition that might reduce the chance of obtaining data required by protocol or that might compromise the ability to give truly informed consent and/or comply with study procedures;
23. Osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures (e.g., tooth extraction, dental implants, oral surgery in the past 6 months), or planned invasive dental procedure during the study; poor oral hygiene, periodontal, and/or pre-existing dental disease;
24. Subject with known hypersensitivity to denosumab or any monoclonal /or polyclonal antibodies or previously received denosumab treatment or to any of the excipients of the IMPs;
25. Known allergies, hypersensitivity, or intolerance to protein-based therapies or to any ingredients (including excipients) of the additional medication (vitamin D, in case replenishment is given) or with a history of any significant drug allergy (e.g., anaphylaxis, hepatotoxicity, immune-mediated thrombocytopenia or anemia) including latex;
26. Corrected serum calcium of < Lower Limit of Normal (LLN) or > ULN at SCR;
27. Individuals with history of tuberculosis or diagnosed with active or latent tuberculosis by interview or interferon-gamma release assay;
28. Vaccinations must be completed 6 weeks prior to dosing in case multiple vaccinations are required and no further vaccinations until the EoS. COVID-19 related vaccinations should not be done within at least 3 weeks prior to SCR and until 3 weeks after dosing. COVID-19 vaccinations should not be done or be planned from 2 days before or on the same day as any ambulatory visits;
29. Participants who smoke more than 10 cigarettes per day or consume equivalent nicotine substitutes, including e-cigarettes or inability to refrain from smoking during the in-house period;
30. Any disease or condition that in the opinion of Investigator, may affect the patient safety or the study results;
31. Subject has a positive test result for SARS-CoV-2 in RT-PCR testing before randomization;
32. Subject has clinical signs and symptoms consistent with COVID-19, e.g., fever, dry cough, dyspnea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 30 days prior to SCR or on admission;
33. Subject who had severe course of COVID-19 (i.e., hospitalization, extracorporeal membrane oxygenation (ECMO), and/or mechanically ventilated);
34. Vulnerable subjects (i.e., persons under any administrative or legal supervision or persons kept in detention);
35. Subjects who are employees of Sponsor, clinical research organization (CRO) or who is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other site staff or relative thereof directly involved in the conduct of the clinical study;
36. Subjects who are not able to read, speak and understand the German language.

Ages: 28 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Day 1 until Day 253
  Area under the concentration-time curve (AUC) from time zero to last quantifiable concentration (AUC0-t)
Cmax | Day 1 until Day 253
  Maximum serum concentration (Cmax)
AUC0-inf | Day 1 until Day 253
  Area under the concentration-time curve (AUC) from time zero to infinity (AUC0-inf) AUC0-inf = AUC from time zero to the last quantifiable concentration (AUC0-t) + last observed concentration (Ct) / terminal rate constant (λz)

SECONDARY OUTCOMES:
tmax | Day 1 until Day 253
  Time corresponding to the occurrence of Cmax (tmax)
t½ | Day 1 until Day 253
  Apparent terminal half-life calculated by ln2/λz (t½)
CL/F | Day 1 until Day 253
  Apparent total body clearance (CL/F)
Vd | Day 1 until Day 253
  Apparent volume of distribution based on the terminal phase (Vd)
λz | Day 1 until Day 253
  Terminal rate constant (λz)
%AUCex | Day 1 until Day 253
  Percentage of AUC0-inf obtained by extrapolation (%AUCex)
Incidence of adverse events (AEs) and serious AEs (SAEs) | Day 1 until Day 253
  Incidence of adverse events (AEs) and serious AEs (SAEs)
blood pressure | Day 1 until Day 253
  supine blood pressure [BP]
pulse rate | Day 1 until Day 253
  pulse rate
body temperature | Day 1 until Day 253
  tympanic body temperature
Clinical laboratory tests | Day 1 until Day 253
  Clinical laboratory tests (hematology, clinical chemistry and urinalysis)
Physical examinations | Day 1 until Day 253
  Physical examinations
Local tolerance | Day 1 until Day 253
  Local tolerance assessed by the Investigator using the Injection site reaction (ISR) Score
Immunogenicity Endpoints | Day 1 until Day 253
  Immunogenicity (ADA and Nab)
AUEC0-t (S-CTX) | Day 1 until Day 253
  Area under S-CTX percent inhibition-time curve from time zero to last quantifiable concentration (AUEC0-t)
AUEC0-16w (S-CTX) | Day 1 until Day 113
  Area under S-CTX percent inhibition-time curve from time zero to Day 113 (i.e., 16 weeks) (AUEC0-16w)
Imax (S-CTX) | Day 1 until Day 253
  Maximum percent inhibition (Imax)
TImax (S-CTX) | Day 1 until Day 253
  Time to reach maximum percent inhibition (TImax)

CONTACTS AND LOCATIONS:
Overall Officials: R Fuhr, MD, Principal Investigator — Parexel
Locations (2):
- Germany (2):
  - Parexel International GmbH, Early Phase Clinical Unit Berlin, Berlin
  - CTC North GmbH & Co KG, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuhr R, Sun X, Wang X, Dong Y, Tai J, Zhou M, Dou C. A three-arm clinical study to compare pharmacokinetic and pharmacodynamic similarity of the denosumab biosimilar LY06006 with reference denosumab in healthy male subjects. Expert Opin Drug Metab Toxicol. 2024 Nov 24:1-9. doi: 10.1080/17425255.2024.2432673. Online ahead of print. PMID 39582128